CLINICAL TRIAL: NCT05698914
Title: Postoperative Telehealth Mindfulness Intervention After Lumbar Spine Surgery: Pilot Randomized Controlled Trial
Brief Title: Telehealth Mindfulness After Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Carrie Brintz, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 221711; K23AT011569 (NIH)
Record Dates: First submitted 2022-12-27; First posted 2023-01-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Spine Surgery; Chronic Low-back Pain; Postsurgical Pain
Keywords: Mindfulness; Telehealth
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are masked to the names and specific details of each intervention arm at time of enrollment, and remain masked to the name and details of the intervention arm to which they are not randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth mindfulness-based intervention (MBI) (Experimental): Eight, weekly telehealth mindfulness sessions delivered one-on-one with mindfulness instructor
  Interventions: Behavioral: Telehealth mindfulness-based intervention (MBI)
- Telehealth Education (EDU) (Active Comparator): Eight, weekly post-surgical educational sessions delivered one-on-one with physical therapist
  Interventions: Behavioral: Telehealth Education

INTERVENTIONS:
Behavioral: Telehealth mindfulness-based intervention (MBI) — The telehealth MBI is adapted from Mindfulness-based cognitive therapy for chronic pain and consists of eight, weekly 75-minute individual sessions (90 minutes allotted for the first session) with a mindfulness interventionist delivering the intervention over telehealth (online with audio and video camera) in addition to the patient receiving their usual postsurgical care. Participants will begin the intervention after completing the 2-week postoperative assessment and within 4 weeks after surgery. Participants will be asked to practice skills between sessions approximately 20-40 minutes per day.
  Arms: Telehealth mindfulness-based intervention (MBI)
Behavioral: Telehealth Education — Participants will receive a written educational booklet at the time of randomization (within 2-4 weeks after surgery) and 8, weekly telehealth sessions lasting 30 minutes in addition to usual postsurgical care. The educational materials are reviewed individually with the participant during weekly telehealth sessions (online with audio and video camera) by a physical therapist.
  Arms: Telehealth Education (EDU)

SUMMARY:
The goal of this pilot clinical trial is to compare two behavioral interventions for patients who are recovering from lumbar spinal surgery for a degenerative spine condition. The study aims to answer the following questions:

1. Is it feasible and acceptable to deliver the interventions and conduct the study procedures in this patient population?
2. Do the interventions benefit patients with regard to pain-related, functional, opioid use, and psychosocial outcomes at 3 and 6 months after surgery, and does one intervention have more benefit than the other?

Participants will be asked to do the following:

1. Complete self-report questionnaires online before spine surgery, and around 2 weeks, 3 months, and 6 months after spine surgery.
2. Complete a sensory pain task before spine surgery, and around 2 weeks, 3 months, and 6 months after spine surgery.
3. Around two weeks after surgery, participants will be randomly assigned by chance to one of two behavioral interventions - Mindfulness or Education. Participants will then be asked to attend 8, weekly sessions with a study treatment coach over telehealth (online with camera and microphone).

DETAILED DESCRIPTION:
This is a pilot randomized clinical trial comparing a telehealth mindfulness-based intervention (MBI) with a telehealth education intervention (EDU) for patients recovering from spine surgery. The procedures will be as follows:

1. Enroll patients prior to lumbar spine surgery for a degenerative spine condition at the Vanderbilt Comprehensive Spine Center. Recruitment, enrollment, and screening will occur at a routine preoperative clinic visit or over the phone.
2. Two weeks after enrolled participants complete surgery, they will be randomized in a 3:2 ratio to either MBI or EDU condition, respectively. Randomization will be stratified by chronic preoperative opioid use (yes/no). The randomization assignments will remain concealed from all study personnel until the time of randomization. The outcome assessor and surgical providers will remain blinded to participant study condition.
3. Within four weeks of surgery, participants will begin the assigned intervention. The interventions will consist of meeting with an interventionist for eight, weekly one-on-one telehealth MBI sessions over an online telehealth platform. MBI sessions will led by a clinical psychologist and will be 75 minutes long (90 minutes for the first session). EDU sessions will be led by a physical therapist and will be 30 minutes long. Sessions will be audio recorded and monitored for fidelity.

3) Participants will complete self-report assessments online prior to surgery, two weeks after surgery (pre-intervention), three months after surgery (post-intervention) and 6 months after surgery.

4) Participants will complete quantitative sensory testing assessments of pain tolerance, pain threshold, and temporal summation of pain prior to surgery, two weeks after surgery, three months after surgery, and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking adults
2. Aged 18 years and older
3. Scheduled for a laminectomy and/or fusion at Vanderbilt Spine Center
4. Scheduled for their first lumbar spine surgery
5. Radiographic evidence of a degenerative condition including but not limited to spinal stenosis, spondylosis with or without myelopathy, and spondylolisthesis
6. Presence of back and/or lower extremity pain persisting for at least 3 months
7. Access to stable internet.
8. Able to participate in weekly, remote sessions with a study therapist for 8 weeks after surgery

Exclusion Criteria:

1. Microsurgical technique as the primary procedure (i.e. isolated laminotomy or microdiscectomy)
2. Having surgery for the primary indication of a spinal deformity
3. Having surgery secondary to pseudarthrosis, trauma, infection, or tumor
4. Current/history of a primary psychotic or major thought disorder or hospitalization for reasons related to psychosis (e.g. Schizophrenia, brief psychotic disorder, delusional disorder). Medication-induced psychosis is not exclusionary.
5. Diagnosis of Alzheimer's disease or another form of dementia
6. Traumatic Brain Injury (greater than mild severity)
7. History of bipolar disorder or dissociative disorder
8. Active substance use disorder (in past month)
9. Current Posttraumatic Stress Disorder (PTSD) symptoms (in past month)
10. Active suicidal ideation with intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Enrollment Rate | Through enrollment completion, approximately 21 months
  Proportion of participants approached who are eligible and enroll in the study
Participant study retention | Through study completion, approximately 28 months
  Proportion of participants who complete the study (6 month assessment)
Session attendance | Through 3 months postoperative
  Average percentage of sessions attended
Intervention Satisfaction | 3 months postoperative
  Proportion of participants reporting overall satisfaction levels greater than or equal to 7 out of 10
Home practice completion | Through 3 months postoperative
  Average days practiced out of days assigned practice (MBI group only)

SECONDARY OUTCOMES:
Pain Bothersomeness | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  One item assessing how bothersome pain has been in the past 7 days from 0 = not at all to 4 = extremely. A lower scores indicates lower pain bothersomeness.
Pain Interference Short-form 8a | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  Pain Interference short-form 8a from the Patient Reported Outcomes Measurement Information System scale. Measures interference of pain over the past 7 days. Consists of 8 items with response options from 1 = not at all to 5 = very much. A lower score indicates lower pain interference, or a better outcome.
Overall Pain Intensity Overall Pain Intensity | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  1 item from the Patient Reported Outcomes Measurement Information System (PROMIS), with average pain intensity over the past 7 days rated on 0-10 scale with lower values indicating less pain, or better outcome.
Back and leg pain intensity | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  2 items assessing back and leg pain intensity on a scale of 0-10 over the past 7 days, described as pain when off medication or medication has worn off. Lower scores indicate less pain, or better outcome.
Self-reported opioid medication use | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  Measured as average number of opioid pills per day (name and dose specified) and converted to morphine equivalent dose.
Opioid medication collected from the Electronic Medical Record | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  Opioid medication prescription from patient's electronic medical record to cross-reference self-reported opioid medication use
Anxiety Short Form 4a | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  Anxiety short-form 4a - Patient Reported Outcomes Measurement Information System. 4 items assessing anxiety symptoms in the past 7 days (e.g. "I felt fearful") with response options from 1 = never to 5 = always. Lower scores represent lower anxiety, a better outcome
Depression Short Form 4a | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  Depression short-form 4a - Patient Reported Outcomes Measurement Information System scale. 4 items assessing depressive symptoms over the past 7 days (e.g. "I felt worthless) with response options from 1 = never to 5 = always. A lower score indicates less depression, a better outcome.
Sleep Disturbance Short Form 4a | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  Sleep disturbance short-form 4a - Patient Reported Outcomes Measurement Information System scale. 4 items assessing sleep disturbance over the past 7 days (e.g. "I had difficulty falling asleep) with response options from 1 = not at all to 5 = very much (1 item reverse-scored). A lower score indicates less sleep disturbance, a better outcome.
Oswestry Disability Index | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  Assesses impact of pain on level of functioning in 10 areas (e.g. walking, sleep, social life) with 10 items with response options with scores 0 to 5. Lower scores indicate lower level of disability due to pain, a better outcome.
Pain Catastrophizing Scale | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  13 items assessing thoughts and feelings when in pain (e.g. "I become afraid that the pain will get worse" with response options ranging from 0 = never to 4 = all the time. Lower scores indicate lower pain catastrophizing, a better outcome.
Pain Self-efficacy Questionnaire | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  10 items assessing confidence in ability to do certain things despite pain (e.g. "I can enjoy things, despite the pain" with response options 0 = not at all to 6 = completely. Higher scores indicate greater pain self-efficacy, a better outcome.
Perceived Stress Scale - 4 | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  4 items assessing perceived level of stress in the past month (e.g. "In the last month, how often have you felt that you were unable to control the important things in your life?"), with response options ranging from 0 = never to 4 = very often (2 items reverse-scored). Lower scores indicate lower perceived stress, a better outcome.
Tampa Scale for Kinesiophobia -13 | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  13 items assessing fear of movement (e.g. "I'm afraid that I might injure myself if I exercise" with response options ranging from 1 = strongly disagree to 4 = strongly agree. Lower scores indicate lower levels of kinesiophobia, a better outcome.
Five Facet Mindfulness Questionnaire - 15 | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  15 items assessing 5 facets of mindfulness, including observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Response options range from 1 = never to 5 = always (7 items reverse scored). Higher scores indicate higher levels of mindfulness, a better outcome.
Pain Tolerance | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  Using an ischemic task involving squeezing a dynamometer followed by inflated blood pressure cuff on arm, the point at which the stimulus (inflated blood pressure cuff) can no longer be tolerated by the participant.
Pain Threshold | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  Using an ischemic task involving squeezing a dynamometer followed by inflated blood pressure cuff on arm, the point at which the stimulus (inflated blood pressure cuff) is first experienced as painful by the participant.
Temporal Summation of Pain Temporal Summation of Pain | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  Using a punctate stimuli (von frey hairs of 100g and 180g of force to the finger), the reported highest pain intensity on a scale of 0 to 100 during repeated brief stimuli at a constant intensity
Physical Function | Preoperative, 2 weeks postoperative, 3 months postoperative, 6 months postoperative
  Physical Function short-form 4a - Patient Reported Outcomes Measurement Information System. 4 items assessing physical function in the past 7 days (e.g. "Are you able to do chores such as vacuuming or yard work?") with response options from 1 = Unable to do to 5 = Without any difficulty. Higher scores represent better physical function, a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Carrie E Brintz, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT05698914/ICF_000.pdf